CLINICAL TRIAL: NCT06701305
Title: A Single and Multiple-Ascending Dose Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Efinopegdutide (MK-6024) in Otherwise Healthy Obese Participants and the Effect of Multiple Doses of Efinopegdutide on the Pharmacokinetics of Acetaminophen
Brief Title: A Study of Efinopegdutide in Healthy Obese Participants (MK-6024-015)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 6024-015; MK-6024-015 (Other: MSD)
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Healthy
MeSH Terms: interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Efinopegdutide (Experimental): Part 1: Participants receive a single subcutaneous (SC) dose of efinopegdutide.
  Interventions: Drug: Efinopegdutide
- Part 1: Placebo (Placebo Comparator): Part 1: Participants receive a single SC dose of placebo.
  Interventions: Drug: Placebo
- Part 2: Efinopegdutide (Experimental): Part 2: Participants receive multiple SC doses of efinopegdutide titrated from Dosage 1, Dosage 2, Dosage 3, Dosage 4, Dosage 5, or Dosage 6. Participants receive a SC dose of efinopegdutide, Dosage 1 on Days 1 and 8; Dosage 2 on Days 15 and 22; Dosage 3 on Days 29, 36, 43 and 50; Dosage 4 on Days 57, 64, 71 and 78; Dosage 5 on Days 85, 92, 99, 106; and Dosage 6 on Days 113, 120, 127, and 134. Participants also receive oral acetaminophen on Day -2, Day 6, 62, and 83.
  Interventions: Drug: Efinopegdutide; Drug: Acetaminophen
- Part 2: Placebo (Placebo Comparator): Part 2: Participants receive multiple SC doses of Placebo titrated from Dosage 1, Dosage 2, Dosage 3, Dosage 4, Dosage 5, or Dosage 6.
  Participants receive a SC dose of Placebo, Dosage 1 on Days 1 and 8; Dosage 2 on Days 15 and 22; Dosage 3 on Days 29, 36, 43 and 50; Dosage 4 on Days 57, 64, 71 and 78; Dosage 5 on Days 85, 92, 99, 106; and Dosage 6 on Days 113, 120, 127, and 134. Participants also receive oral acetaminophen on Day -2, Day 6, 62, and 83.
  Interventions: Drug: Placebo; Drug: Acetaminophen

INTERVENTIONS:
Drug: Efinopegdutide — Subcutaneous injectable solution
  Other Names: MK-6024
  Arms: Part 1: Efinopegdutide; Part 2: Efinopegdutide
Drug: Placebo — Subcutaneous injectable solution
  Arms: Part 1: Placebo; Part 2: Placebo
Drug: Acetaminophen — Oral solution
  Arms: Part 2: Efinopegdutide; Part 2: Placebo

SUMMARY:
The goal of this study is to learn about the safety of efinopegdutide (MK-6024) and how well overweight healthy people tolerate it. Researchers also want to know what happens to efinopegdutide in a person's body over time when taken as a single dose (Part 1) or as multiple doses (Part 2). In addition, the study will assess the amount of acetaminophen in the blood after receiving different strength doses of efinopegdutide (Part 2 only).

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Is in good health
* Has body mass index (BMI) between 29 kg/m^2 and 38 kg/m^2

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History of clinically significant endocrine, gastrointestinal (GI), cardiovascular (CV), hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* History of cancer (malignancy)
* Positive test(s) for Hepatitis B surface antigen (HBsAg), hepatitis C antibodies, or Human immunodeficiency virus (HIV)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2025-02-18 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 35 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Part 1: Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 35 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.
Part 1: Maximum Plasma Concentration (Cmax) of Efinopegdutide | Pre-dose and at designated time points up to 35 days post dose
  Blood samples will be collected to determine the Cmax of Efinopegdutide.
Part 1: Time to Maximum Plasma Concentration (Tmax) of Efinopegdutide | Pre-dose and at designated time points up to 35 days post dose
  Blood samples will be collected to determine the Tmax of Efinopegdutide.
Part 1: Area Under the Concentration-Time Curve from Time 0 to Last Measurable Concentration (AUC0-last) of Efinopegdutide | Pre-dose and at designated time points up to 35 days post dose
  Blood samples will be collected to determine the AUC0-last of Efinopegdutide.
Part 1: Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of Efinopegdutide | Pre-dose and at designated time points up to 35 days post dose
  Blood samples will be collected to determine the AUC0-Inf of Efinopegdutide.
Part 1: Apparent Terminal Half-life (t1/2) of Efinopegdutide | Pre-dose and at designated time points up to 35 days post dose
  Blood samples will be collected to determine the t1/2 of Efinopegdutide.
Part 1: Apparent Clearance (CL/F) of Efinopegdutide | Pre-dose and at designated time points up to 35 days post dose
  Blood samples will be collected to determine the CL/F of Efinopegdutide.
Part 1: Apparent volume of distribution during terminal phase (Vz/F) of Efinopegdutide | Pre-dose and at designated time points up to 35 days post dose
  Blood samples will be collected to determine the Vz/F of Efinopegdutide.
Part 2: Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 184 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Part 2: Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 184 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.
Part 2: Cmax of Efinopegdutide | At designated time points up to approximately 184 days
  Blood samples will be collected to determine the Cmax of Efinopegdutide.
Part 2: Tmax of Efinopegdutide | At designated time points up to approximately 184 days
  Blood samples will be collected to determine the Tmax of Efinopegdutide.
Part 2: Area Under the Concentration-Time Curve from Time 0 to the End of the Dosing Interval (AUC0-tau) of Efinopegdutide | At designated time points up to approximately 184 days
  Blood samples will be collected to determine the AUC0-tau of Efinopegdutide.
Part 2: t1/2 of Efinopegdutide | At designated time points up to approximately 184 days
  Blood samples will be collected to determine the CL/F of Efinopegdutide.
Part 2: Vz/F of Efinopegdutide | At designated time points up to approximately 184 days
  Blood samples will be collected to determine the Vz/F of Efinopegdutide.
Part 2: Concentration Immediately Before the Next Dose is Administered (Ctrough) of Efinopegdutide | At designated time points up to approximately 184 days
  Blood samples will be collected to determine the Ctrough of Efinopegdutide.

SECONDARY OUTCOMES:
Part 2: AUC0-Inf of Acetaminophen | At designated time points up to approximately 184 days
  Blood samples will be collected to determine the AUC0-inf of Acetaminophen.
Part 2: Cmax of Acetaminophen | At designated time points up to approximately 184 days
  Blood samples will be collected to determine the Cmax of Acetaminophen.
Part 2: Tmax of Acetaminophen | At designated time points up to approximately 184 days
  Blood samples will be collected to determine the Tmax of Acetaminophen.
Part 2: t1/2 of Acetaminophen | At designated time points up to approximately 184 days
  Blood samples will be collected to determine the t1/2 of Acetaminophen.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- QPS-MRA, LLC (Site 0001), South Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com